CLINICAL TRIAL: NCT05342272
Title: Comparison of Gum® HydralTM Moisturizing Gel and Biotene® Oral Gel in Dry Mouth Sensation Reduction: a Randomized Clinical Trial
Brief Title: Comparison of Gum® HydralTM Moisturizing Gel and Biotene® Oral Gel in Dry Mouth Sensation Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Sunstar Suisse (Unknown)
Responsible Party: Principal Investigator, Domenico Dalessandri, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NP2789
Record Dates: First submitted 2021-11-27; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Xerostomia
Keywords: Surveys and Questionnaires
MeSH Terms: conditions — Xerostomia | interventions — Xylitol; Lactoperoxidase; Muramidase; Lactoferrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GUM Hydral Moisturizing Gel (Experimental): One group of 20 patients receiving GUM® Hydral® Moisturizing Gel (test group): they were be instructed to apply during a 28 days treatment period 1 to 2 cm of gel to gums, oral mucosa membrane and tongue, repeating as many times as necessary.
  Interventions: Drug: Betaine taurine PVP gel
- Biotene Oral Balance Gel (Active Comparator): One group of 20 patients receiving Biotene® Oral Balance Gel (control group): they were be instructed to apply during a 28 days treatment period 1 to 2 cm of gel to gums, oral mucosa membrane and tongue, repeating as many times as necessary.
  Interventions: Drug: Xylitol, Lactoperoxidase, Lysozyme, Lactoferrin

INTERVENTIONS:
Drug: Betaine taurine PVP gel — At the beginning of the trial (t0) each patient received a print-out summarizing the instructions for use of the products: they were instructed to apply during a 28 days treatment period 1 to 2 cm of GUM Hydral® gel to gums, oral mucosa membrane and tongue, repeating as many times as necessary, and to brush their teeth with GUM® Technique® Pro soft compact toothbrush (Sunstar Europe S.A., Etoy, Switzerland) using GUM® Hydral® Toothpaste (Sunstar Europe S.A., Etoy, Switzerland) at least twice a day. The first application was done by the participants themselves under the supervision of the same operator that provided them both oral and written usage instructions. They had to refrain from using any other commercial mouthrinse, toothpaste or saliva supplements during the trial.
  Other Names: GUM Hydral® Gel
  Arms: GUM Hydral Moisturizing Gel
Drug: Xylitol, Lactoperoxidase, Lysozyme, Lactoferrin — At the beginning of the trial (t0) each patient received a print-out summarizing the instructions for use of the products: they were instructed to apply during a 28 days treatment period 1 to 2 cm of Biotene® Oral Balance gel to gums, oral mucosa membrane and tongue, repeating as many times as necessary, and to brush their teeth with GUM® Technique® Pro soft compact toothbrush (Sunstar Europe S.A., Etoy, Switzerland) using GUM® Hydral® Toothpaste (Sunstar Europe S.A., Etoy, Switzerland) at least twice a day. The first application was done by the participants themselves under the supervision of the same operator that provided them both oral and written usage instructions. They had to refrain from using any other commercial mouthrinse, toothpaste or saliva supplements during the trial.
  Other Names: Biotene® Oral Balance Gel
  Arms: Biotene Oral Balance Gel

SUMMARY:
Background. Xerostomia is estimated to affect up to 50% of the adult population and especially the elderly suffer from dry mouth sensation. Our aim was to compare the efficacy of GUM® Hydral® Moisturizing Gel and Biotene® Oral Balance Gel in dry mouth sensation reduction.

Study design and Methods. Forty patients, reporting dry mouth sensation between 4 to 10 on a 0 (no discomfort) to 10 (extreme discomfort) scale, were divided in two parallel groups respectively treated with GUM® Hydral® and Biotene® Gel following a stratified randomization list (t0). Patients and the research assistants were blinded to group assignment. Patients underwent measurements of unstimulated and stimulated whole saliva flow and weekly (t1, t2, t3, t4) were asked to fill in a patient questionnaire and daily a journal to evaluate the dry mouth symptoms and the subjective perception of changes in the symptoms during one month of treatment. After data collection (t1-t4), patients were medically followed over the next six months in order to detect any long-term side effects (t5).

DETAILED DESCRIPTION:
After clinical history analysis subjects were randomized, using a stratified randomization list which considered as main prognostic factor the presence of a systemic pathology/drug assumption responsible for the onset of xerostomia, into 2 parallel groups: one group of 20 patients receiving GUM® Hydral® Moisturizing Gel (test group); one group of 20 patients receiving Biotene® Oral Balance Gel (control group).

In order to guarantee the allocation concealment, the randomization list was prepared after patient inclusion in the study by a centralized office, responsible for the integrity of the whole randomization protocol, and after that treatment products presented in kits were distributed to each patient. Blinding of the evaluators and patients was obtained using the same white anonymous packages for both tested products. The stratification was obtained separating the patients in two groups, with and without the presence of a systemic pathology/drug assumption responsible for the xerostomia onset, and then generating two separated randomized lists.

At the beginning of the trial (t0) each patient received a print-out summarizing the instructions for use of the products: they were instructed to apply during a 28 days treatment period 1 to 2 cm of gel to gums, oral mucosa membrane and tongue, repeating as many times as necessary, and to brush their teeth with GUM® Technique® Pro soft compact toothbrush (Sunstar Europe S.A., Etoy, Switzerland) using GUM® Hydral® Toothpaste (Sunstar Europe S.A., Etoy, Switzerland) at least twice a day. The first application was done by the participants themselves under the supervision of the same operator that provided them both oral and written usage instructions. They had to refrain from using any other commercial mouthrinse, toothpaste or saliva supplements during the trial and they were asked to complete a "patient questionnaire" at the same time of the day (in the morning, at the hospital prior to their clinical examination) at t0, t1 (after 1st week), t2 (2nd week), t3 (3rd week) and at the end of the trial, t4 (4th week), and a "daily journal".

The "patient questionnaire" was used to record the severity of the dry mouth sensation and changes in the symptoms (thanks to a VAS scale and dichotomous variables). It also contained questions to evaluate the quality of life (QoL) improvement (psychological impact and social well-being), the convenience of use and overall feeling (at t4), and the organoleptic properties of the tested products.

In the "daily journal", patients indicated on a dedicated calendar the times of product use, they reported their subjective sensation of oral dryness 3 times a day (morning, around 12 AM - 2 PM, evening) on a Visual Analogue Scale (VAS) ranging from 0 (well lubricated mouth) to 10 (worst possible dry mouth feeling), and they answered the following two questions (once a day at the same time): "How many minutes after the use of the gel did you feel dry mouth relief?" and "How long (expressed in minutes) did the dry mouth relief last (after the use of the gel)?" to record the perceived speed and duration of effects of the products and their pleasantness of use.

The salivary flow rate is the amount of saliva produced by salivary glands in the time unit and it can be divided into unstimulated (which is independent of the presence of stimuli as food and chewing) and stimulated (secreted in response to sensory stimulation, gustatory and masticatory mainly)40.

At t0, after one hour of abstinence from drinking, eating and smoking, the patients were characterized by means of an unstimulated (Whole Resting Saliva - WRS) and a stimulated (Whole Stimulated Saliva - WSS) whole saliva flow determination using the spitting method between 11.00 and 12.00 a.m. under controlled temperature and humidity conditions37,39,40,41. WRS was determined collecting saliva produced during a time span of 5 minutes37; subsequently, WSS was determined collecting saliva produced during a time span of 1 minute, after 5 minutes chewing a paraffin soft ball.

The enrolled subjects were submitted to a rigid protocol of behavioral norms in preparation for salivary collection37,38,39,40,41. Patients were advised to keep a relaxed attitude and not to practice sports and/or physical efforts in the two days prior to the salivary collection37,41. On the sampling day, participants had to be free from symptoms of fever and/or cold; if they were hungry or thirsty, they could eat or drink water, but immediately afterwards they had to brush their teeth with a provided toothpaste37. During the collection periods, subjects remained comfortably seated and swallowed residual saliva present in the mouth before the beginning of tests37. Then, with the head down and the mouth slightly open, saliva was allowed to drip from the lower lip into a pre-weight, dry, deionized and sterilized plastic test tube37.

At t0, t1, t2, t3, and t4 the same operator, blind regarding patient treatment group assignment, completed the ROAG (Revised Oral Assessment Guide) scale and reported any local irritation or allergic reaction caused by the product. In case of changes in medication assumption changes during the study period, patients were excluded from the sample.

After the conclusion of the data collection, patients were medically followed in the subsequent six months in order to recognize any long-term side effect appearance (t5).

ELIGIBILITY:
Inclusion Criteria:

* Use of a dry mouth product in the past 6 months
* Level of discomfort from dry mouth between 4 to 10 on a 0 (no discomfort) to 10 (extreme discomfort) scale
* Use of a dry mouth product at least 2-3 times per week

Exclusion Criteria:

* History of any treatment for cancer in the last 3 months
* Recurrence of cancer and end stage of it
* Being on a restrictive dietary regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Dry mouth sensation relief change | Beginning, after 1 - 2 - 3 - 4 weeks, after 6 months
  Patients were asked to complete a "patient questionnaire" at the same time of the day at t0, t1 (after 1st week), t2 (2nd week), t3 (3rd week) and at the end of the trial, t4 (4th week), and a "daily journal". The "patient questionnaire" was used to record the severity of the dry mouth sensation and changes in the symptoms (thanks to a VAS scale and dichotomous variables). In the "daily journal", patients indicated on a dedicated calendar the times of product use, they reported their subjective sensation of oral dryness 3 times a day on a Visual Analogue Scale (VAS) ranging from 0 (well lubricated mouth) to 10 (worst possible dry mouth feeling), and they answered the following two questions: "How many minutes after the use of the gel did you feel dry mouth relief?" and "How long (expressed in minutes) did the dry mouth relief last (after the use of the gel)?" to record the perceived speed and duration of effects of the products and their pleasantness of use.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Dalessandri, Prof., Principal Investigator — Università degli Studi di Brescia
Locations (2):
- Italy (2):
  - ASST Spedali Civili di Brescia, Brescia, BS
  - ASST Spedali Civili di Brescia, Brescia

IPD SHARING:
Plan to Share IPD: No